CLINICAL TRIAL: NCT02869243
Title: A Dose Escalation Phase I Study Of Human- Recombinant Bone Morphogenetic Protein 4 Administrated Via Convection-Enhanced Delivery In Patients With Progressive And/Or Multiple Recurrent Glioblastoma Multiforme
Brief Title: A Dose Escalation Phase I Study Of Human- Recombinant Bone Morphogenetic Protein 4 Administrated Via CED In GBM Patients
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Stemgen (Industry)
Collaborators: ORION Clinical Services (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: hrBMP4-001
Record Dates: First submitted 2016-08-02; First posted 2016-08-16 (Estimated); Last update posted 2024-02-16 (Actual); Status verified 2024-02

CONDITIONS: Glioblastoma
Keywords: A malignant growing astrocytoma of central nervous system
MeSH Terms: conditions — Glioblastoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- hrBMP4 (Experimental): Intra-tumour and interstitial convection enhanced delivery (CED) as a continuous infusion via intracranial catheters of hrBMP4 solution and gadolinium
  Interventions: Drug: hrBMP4

INTERVENTIONS:
Drug: hrBMP4 — Patients will undergo a resection or biopsy of the tumour, confirmation of viable malignant glioma tumour cells and intratumour/interstitial placement under neuronavigational guidance of 2 or 3 catheters.
  Catheters will be placed during a second procedure a few days later based upon the patient's condition.
  Patients will receive intra-tumour and interstitial CED of increasing amounts of hrBMP4 solutions (starting dose of 0.5 mg) and 1:70 gadolinium-diethylenetriamine pentaacetic acid (Gd-DTPA) in a total of 44-66ml over up to 4-6 days. Gd-DTPA will be co-infused with BMP4 to determine the extent of intra-tumour and interstitial drug delivery. HrBMP4 will be delivered as a continuous infusion via the intracranial catheters.
  Other Names: Recombinant Bone Morphogenic Protein-4; Device:Intracranial Catheter

SUMMARY:
The purpose of the study is to evaluate the feasibility and safety of intra-tumor and interstitial therapy with hBMP4 in increasing doses in patients with progressive and/or multiple recurrent Glioblastoma multiforme (GBM).

DETAILED DESCRIPTION:
This multicentre, open-label, dose escalating, Phase I study will enrol approximately 18 patients with progressive and/or multiple recurrent GBM, who after failure of standard therapies will receive GMP Human- recombinant Bone Morphogenetic Protein 4 via intra-tumour and interstitial delivery by CED.

Patients will undergo a resection or biopsy of the tumour, confirmation of viable malignant glioma tumour cells during frozen section performed by the institutional pathologists, and intra-tumor and interstitial placement under neuronavigational guidance of 2 or 3 catheters. No catheters will be placed at time of resection. After resection, catheters will be placed during a separate procedure several days later based upon the patient's condition as determined by both a clinical examination and routine MRI scan.

Patients will receive intra-tumour and interstitial CED of increasing amounts of hrBMP4 solutions (at a starting dose of 0.5 mg) and 1:70 gadolinium-diethylenetriamine pentaacetic acid (Gd-DTPA) in a total of 44-66 ml over up to 4-6 days at the discretion of the investigator.

Gd-DTPA will be co-infused with hrBMP4 to determine the extent of intra-tumour and interstitial drug delivery. Patients will be hospitalized from the time of the original surgery until the end of infusion of hrBMP4.

Patients will be followed for the duration of the study. The primary endpoint of the study is monitoring feasibility and patient safety for the incidence of Dose-Limiting Toxicity (DLT) following intra-tumour and interstitial therapy with hrBMP4 and to determine whether there is a Maximum Tolerated Dose (MTD).

ELIGIBILITY:
Inclusion Criteria:

To be eligible for inclusion into this study, each patient must fulfil the following inclusion criteria ≤ 28 days prior to the anticipated surgery date:

1. Malignant glioma (WHO grade III or IV) who have undergone conventional treatment, including surgery (gross total resection or unintentional partial resection with residual tumour) or biopsy (with residual tumour), and/or radiation therapy, and/or chemotherapy, and/or Temozolomide and have progressive and/or multiple recurrent GBM. Preoperative assessment by clinical presentation and CT/MRI appearance of the lesion will identify suitable candidates.
2. Age 18-75 years.
3. Karnofsky >70 (see APPENDIX C: EXAMPLE OF PERFORMANCE STATUS: KARNOFSKY SCALE).
4. Stable dose of corticosteroids no longer than 4 weeks prior to enrolment.
5. Females of childbearing potential must have a negative serum or urine pregnancy test.

   Females who have undergone surgical sterilization or who have been postmenopausal for at least 2 years are not considered to be of childbearing potential.
6. Females of childbearing potential and males who have not undergone surgical sterilization must agree to practice a form of effective contraception prior to entry into the study and for 1 month after the end of infusion.

   Effective contraception:

   If female, is non-lactating, has a negative urine pregnancy test result, and does not plan on becoming pregnant during the study, or not of childbearing potential (hysterectomy or tubal ligation at least 6 months prior to entry to the study or post-menopausal for 1 year); if of childbearing potential (including peri-menopausal women who have had a menstrual period within one year) must practice or be willing to continue to practice acceptable birth control from screening and until 1 month after the study medication has been discontinued.

   Acceptable birth control includes:
   1. Combined (oestrogen and progestogen containing) hormonal contraception;
   2. Associated with inhibition of ovulation; oral OR intravaginal OR transdermal;
   3. Progestogen-only hormonal contraception associated with inhibition of ovulation: oral OR injectable OR implantable;
   4. Progestogen-only oral hormonal contraception, where inhibition of ovulation is not the primary mode of action;
   5. Intrauterine device (IUD);
   6. Intrauterine hormone-releasing system (IUS);
   7. Bilateral tubal occlusion;
   8. Vasectomised partner;
   9. Sexual abstinence;
   10. Male or female condom with or without spermicide;
   11. Cap, diaphragm or sponge with spermicide. Complies with The Heads of Medicines Agencies (HMA) Recommendations Related to Contraception and Pregnancy Testing in Clinical Trials (Sept 2014).

   The definition of effective contraception will be based on the judgment of the investigator.
7. Ability to understand and the willingness to sign a written informed consent document.

Exclusion Criteria:

To be eligible for inclusion into this study, each patient must violate none of the following exclusion criteria ≤ 28 days prior to the anticipated surgery date:

1. Patients who had chemotherapy, radiotherapy or other anti-neoplastic therapy (within 4 weeks or 5x half-life whichever is shorter) prior to study treatment or those who have not recovered to Grade ≤1 or returned to baseline from any acute treatment-related toxicities of the previous therapy except for alopecia and Grade 2 neuropathy.
2. Patients who are receiving any other investigational agents.
3. Life expectancy <3 months
4. Haematological dysfunction defined as:

   * White blood cell (WBC) count <3.0 x 109/L;
   * Absolute neutrophil count <1.5 x 109/L;
   * Haemoglobin level <10.0 g/dL;
   * Platelet count <100 x 109/L.
5. Liver dysfunction defined as:

   * Aspartate transaminase (AST) >2.5 x the upper limit of normal (ULN) for age and gender;
   * Alanine transaminase (ALT) >2.5 x the ULN for age and gender;
   * Bilirubin >1.5 x the ULN for age and gender.
6. Renal dysfunction defined as:

   - Creatinine clearance <60 mL/min/1.73 m2 for patients with creatinine levels above institutional normal for age and gender.
7. Serology indicating active infection with Hepatitis B or C, or HIV.
8. Significant co-morbidity, including coagulation disorders.
9. Pregnancy or unwillingness to practice reliable birth control.
10. Presence of another active malignancy less than 2 years previously (exception: non-melanoma skin cancer).
11. Multifocal, bilateral
12. Midline shift more than 5 mm

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2017-07-18 (Actual); Primary Completion 2020-10-16 (Actual); Study Completion 2021-06-30 (Actual)

PRIMARY OUTCOMES:
DLTs | Up to 8 Weeks after each cohort of 3 patients
  Number of patients who experienced Dose-Limiting Toxicities. DLT is collected to determine Maximum-Tolerated Dose (MTD)

SECONDARY OUTCOMES:
Tumor response | Within 28 days before resection, intraoperative, up to 24 hours post start infusion, after 4-6 days post start infusion (end of infusion) and 4, 12, 24, 36, 48 and 52 weeks after hospitalization
  MRI scans with the following variables: volumetric T1, T2, volumetric Fluid Attenuated Inversion Recovery (FLAIR) and volumetric T1 with contrast. Preoperative assessment by clinical presentation and MRI appearance of the tumour burden will be taken and will be used as the reference point to determine the objective tumour response.
  Objective tumour response: Duplicates of all scans are to be made at the time of each scan and to be retained for the option of a central reading at the end of the trial. Tumour responses must be confirmed by repeat evaluations which should be performed no less than 4 weeks after the criteria of response was first met.
  Tumor response will be evaluated in accordance to Macdonald criteria
EORTC QLQ-C30 Summary Score | After 4-6 days post start infusion (end of infusion) and during 4,8,12 and 52 weeks after hospitalization
  The EORTC quality of life questionnaire (QLQ-C30) will be used to assess quality of life.
  The questionnaires will be available in local languages as per country requirements.
Maximum observed plasma concentration of BMP4 (Cmax) | Prior to the infusion, after 4-6 days post start infusion (end of infusion) and 4 weeks after hospitalization
  Blood samples were obtained and plasma concentrations were determined using a validated high-pressure liquid chromatography method.
Lowest concentration of BMP4 in the blood (Ctrough) | Prior to the infusion, after 4-6 days post start infusion (end of infusion) and 4 weeks after hospitalization
  Blood samples were obtained and plasma concentrations were determined using a validated high-pressure liquid chromatography method.
Area under the curve (AUC∞) | Prior to the infusion, after 4-6 days post start infusion (end of infusion) and 4 weeks after hospitalization
  Blood samples were obtained and plasma concentrations were determined using a validated high-pressure liquid chromatography method.
Central and peripheral volumes of distribution (Vd) | Prior to the infusion, after 4-6 days post start infusion (end of infusion) and 4 weeks after hospitalization
  Blood samples were obtained and plasma concentrations were determined using a validated high-pressure liquid chromatography method.
Clearance | Prior to the infusion, after 4-6 days post start infusion (end of infusion) and 4 weeks after hospitalization
  Blood samples were obtained and plasma concentrations were determined using a validated high-pressure liquid chromatography method.
Half-life (t1/2) | Prior to the infusion, after 4-6 days post start infusion (end of infusion) and 4 weeks after hospitalization
  Blood samples were obtained and plasma concentrations were determined using a validated high-pressure liquid chromatography method.

CONTACTS AND LOCATIONS:
Overall Officials: Francesco DiMeco, PI, Principal Investigator — Istituto Neurologico C. Besta Milan Italy
Locations (4):
- Tel Aviv Sourasky Medical Center, Tel Aviv, Israel
- Istituto Neurologico Carlo Besta, Milan, Italy
- Netherlands (2):
  - VU University Medical Center, Amsterdam
  - Erasmus University Medical Center, Department of Neurosurgery, Rotterdam

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Bos EM, Binda E, Verploegh ISC, Wembacher E, Hoefnagel D, Balvers RK, Korporaal AL, Conidi A, Warnert EAH, Trivieri N, Visioli A, Zaccarini P, Caiola L, van Wijck R, van der Spek P, Huylebroeck D, Leenstra S, Lamfers MLM, Ram Z, Westphal M, Noske D, Legnani F, DiMeco F, Vescovi AL, Dirven CMF. Local delivery of hrBMP4 as an anticancer therapy in patients with recurrent glioblastoma: a first-in-human phase 1 dose escalation trial. Mol Cancer. 2023 Aug 10;22(1):129. doi: 10.1186/s12943-023-01835-6. PMID 37563568